CLINICAL TRIAL: NCT02381964
Title: Pilot, Randomized, Placebo-controlled, Double-blind, 3-arm Parallel Groups Trial in Healthy Females to Assess Cerebral Haemodynamics and Energy Expenditure During Cognitive Performance After Supplementation With Two Different Multivitamin / Mineral Preparations.
Brief Title: The Effects of Differing Cognitive Task Demands on Whole-body Energy Metabolism and Cerebral Blood-flow: Modulation by Multivitamins/Minerals and Coenzyme Q10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, David Kennedy, Professor David Kennedy, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 9L4
Record Dates: First submitted 2015-02-12; First posted 2015-03-06 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Metabolic Processes
Keywords: cerebral blood flow; cognitive function; vitamins; energy expenditure; NIRS; Indirect calorimetry
MeSH Terms: interventions — Supradyn

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Dietary Supplement: Placebo
- 1RDA+CoQ10 (Experimental): Supradyn® (1RDA+CoQ10) containing vitamins and minerals at levels up to 100% of the 2008 European Union recommended dietary allowances (RDAs), plus 4.5 mg CoQ10 (1RDA+CoQ10).
  Interventions: Dietary Supplement: Supradyn® (1RDA+CoQ10)
- 3RDA (Experimental): Supradyn® (3RDA) containing vitamins and minerals at levels up to 300% of the 1990 European Union RDAs (3RDA).
  Interventions: Dietary Supplement: Supradyn® (3RDA)

INTERVENTIONS:
Dietary Supplement: Supradyn® (1RDA+CoQ10)
  Arms: 1RDA+CoQ10
Dietary Supplement: Supradyn® (3RDA)
  Arms: 3RDA
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
When completing difficult tasks, the brain requires faster delivery of energy sources (oxygen and glucose) via the blood. There is evidence to suggest that some nutritional supplements may increase blood circulation in the brain which can result in improved task performance. The purpose of the study is to evaluate the effects of a multivitamin/mineral preparation (containing a range of vitamins and minerals as contained in commonly consumed multivitamin/minerals available off the shelf) in healthy females on cerebral (brain) blood flow and energy expenditure during cognitive task performance.

DETAILED DESCRIPTION:
Vitamins, minerals and CoQ10, exert a number of physiological effects directly relevant to energy supply and metabolism. Therefore it is hypothesized that the nutritional interventions in this trial will facilitate brain metabolic substrate distribution and utilisation during demanding brain activities with a potential benefit on task performance. This pilot, double-blind, placebo controlled, 3-arm parallel groups trial will utilise two concomitant non-invasive techniques:

* Near Infrared Spectroscopy (NIRS) and
* Indirect Calorimetry (ICa). The NIRS will be utilised to measure the rate of delivery of metabolic substrates (via cerebral blood flow i.e. concentrations of total-haemoglobin) and oxygen extraction from the blood (concentration of deoxy-haemoglobin) in the frontal cortex of the brain during cognitive tasks.

The ICa calculated from exhaled gas analysis will be utilised to quantify the overall 'energy' costs of performance of tasks in terms of oxygen uptake, carbon dioxide production, energy expenditure, and substrate (fat and carbohydrate) metabolism.

Cognitive tasks of differing levels of difficulty will be utilised with the hypothesis that energy expenditure parameters and blood flow/oxygen extraction will increase with rising task demands, and that any treatment related effect will be more evident under conditions of increased neural activity. The effects on the above mentioned parameters of two multivitamin/multimineral preparations (MMP) will be compared to placebo subsequent to single dose administration (acute) and following daily administration over an eight week period (chronic). The nutritional interventions are expected to improve nutritional status and thereby facilitate energy supply and metabolism and to have positive impact on the study parameters. The effects of the nutritional interventions on nutritional status will be evaluated by measuring the plasma/serum concentrations of a selected subset of analytes. It is hypothesized that the nutritional status at baseline and after eight week supplementation period will have an impact on metabolic substrate conversion, oxygen utilisation, cerebral blood flow and cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

Healthy females aged 25 to 50 years.

* Female subjects of childbearing potential must be using a medically acceptable form of birth control and have a negative pregnancy test at screening.
* Subjects agree to abstain throughout the trial from intake of MMP or supplements containing CoQ10.
* Body mass index (BMI) in the range of 18.50-34.99 kg/m2 (extremes included; including normal weight, overweight and class I obese subjects according to WHO BMI classification (WHO 2004)).
* Subjects are, in the opinion of the investigator willing to participate in all scheduled visits, to adhere to the treatment plan, and other trial procedures according to the protocol.
* Subjects accept to refrain from alcohol intake 24 hours and to fast 12 hours before the visits.
* Subjects do not have any condition which may interfere with the subject's ability to perform assessments (i.e. colour blindness) and successfully completes training
* Subjects provide a personally signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the trial and understood and accepts these.

Exclusion Criteria:

Physical parameters (including vital signs, e.g., blood pressure, pulse rate, respiratory rate and body temperature) deviating from normal and with clinical relevance.

* Acute infection at screening or randomization.
* A history of, neurological or psychiatric diseases excluding anxiety or depression.
* Current diagnosis of depression or anxiety.
* A history or current diagnosis of diseases, for which use of MMP might be contraindicated or utilisation of MMP might be affected (e.g., iron accumulation, iron utilisation disorders, hypercalcemia, hypercalciuria, impaired renal function, hypervitaminosis A, hypervitaminosis D).
* A history of significant head trauma.
* Smoker (smoking within the last 3 months).
* Excessive use of caffeine (> 500 mg caffeine per day) from all dietary sources.
* History of migraines within the last five years.
* Current intake of pharmaceuticals (with exception of oral contraceptives, or other routine medications to treat benign conditions, such as antibiotics to treat acne).
* Habitual intake of MMP and dietary supplements within the last 4 weeks (defined as ≥3 consecutive days or ≥4 days in total per week).
* Current or history of drug or alcohol abuse in the opinion of the investigator.
* Current pregnancy or lactation.
* Participation in another clinical trial within 30 days prior to screening.
* Any condition which may interfere with the subject's ability to perform assessments (i.e. colour blindness).
* Any history of hypersensitivity to the investigational medicinal product or its active or inactive constituents or any food allergy or intolerance.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Concentration change in oxygenated hemoglobin (Near Infrared Spectroscopy) | 1 hour post dose
Fat oxidation (Indirect calorimetry) | 1 hour post dose
Concentration change in deoxygenated hemoglobin (Near Infrared Spectroscopy) | 1 hour post dose
Concentration change in total hemoglobin (Near Infrared Spectroscopy) | 1 hour post dose
Concentration change in oxygenated hemoglobin (Near Infrared Spectroscopy) | 56 days post dose
Concentration change in deoxygenated hemoglobin (Near Infrared Spectroscopy) | 56 days post dose
Concentration change in total hemoglobin (Near Infrared Spectroscopy) | 56 days post dose
Carbohydrate oxidation (Indirect calorimetry) | 1 hour post dose
Total energy expenditure (Indirect calorimetry) | 1 hour post dose
Fat oxidation (Indirect calorimetry) | 56 days post dose
Carbohydrate oxidation (Indirect calorimetry) | 56 days post dose
Total energy expenditure (Indirect calorimetry) | 56 days post dose

SECONDARY OUTCOMES:
Serial 3 subtractions accuracy (Computerised cognitive task) | 1 hour post dose
Serial 3 subtractions accuracy (Computerised cognitive task) | 56 days post dose
Serial 7 subtractions accuracy (Computerised cognitive task) | 1 hour post dose
Serial 7 subtractions accuracy (Computerised cognitive task) | 56 days post dose
Serial 17 subtractions accuracy (Computerised cognitive task) | 1 hour post dose
Serial 17 subtractions accuracy (Computerised cognitive task) | 56 days post dose
3-back task accuracy (Computerised cognitive task) | 1 hour post dose
3-back task reaction time (Computerised cognitive task) | 1 hour post dose
3-back task accuracy (Computerised cognitive task) | 56 days post dose
3-back task reaction time (Computerised cognitive task) | 56 days post dose
Stroop task accuracy (Computerised cognitive task) | 1 hour post dose
Stroop task reaction time (Computerised cognitive task) | 1 hour post dose
Stroop task accuracy (Computerised cognitive task) | 56 days post dose
Stroop task reaction time (Computerised cognitive task) | 56 days post dose
Subjective rating of task difficulty for Serial 3 subtractions (Computerised Visual Analogue Scale) | 1 hour post dose
Subjective rating of task difficulty for Serial 7 substractions (Computerised Visual Analogue Scale) | 1 hour post dose
Subjective rating of task difficulty for Serial 17 substractions (Computerised Visual Analogue Scale) | 1 hour post dose
Subjective rating of task difficulty for 3 back task (Computerised Visual Analogue Scale) | 1 hour post dose
Subjective rating of task difficulty for stroop task (Computerised Visual Analogue Scale) | 1 hour post dose
Subjective rating of task difficulty for Serial 3 subtractions (Computerised Visual Analogue Scale) | 56 days post dose
Subjective rating of task difficulty for Serial 7 subtractions (Computerised Visual Analogue Scale) | 56 days post dose
Subjective rating of task difficulty for Serial 17 subtractions (Computerised Visual Analogue Scale) | 56 days post dose
Subjective rating of task difficulty for 3 back task (Computerised Visual Analogue Scale) | 56 days post dose
Subjective rating of task difficulty for stroop task (Computerised Visual Analogue Scale) | 56 days post dose
Subject ratings of energy levels (Computerised Visual Analogue Scale) | 1 hour post dose
Subject ratings of energy levels (Computerised Visual Analogue Scale) | 56 days post dose
Subject ratings of calmness (Computerised Bond-Lader mood scales) | 1 hour post dose
Subject ratings of calmness (Computerised Bond-Lader mood scales) | 56 days post dose
Subject ratings of contentedness (Computerised Bond-Lader mood scales) | 1 hour post dose
Subject ratings of contentedness (Computerised Bond-Lader mood scales) | 56 days post dose
Subject ratings of alertness (Computerised Bond-Lader mood scales) | 1 hour post dose
Subject ratings of alertness (Computerised Bond-Lader mood scales) | 56 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: David O Kennedy, PhD, Principal Investigator — Northumbria University
Locations (1):
- Brain performance and nutrition research centre, Northumbria university, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Derived] Kennedy DO, Stevenson EJ, Jackson PA, Dunn S, Wishart K, Bieri G, Barella L, Carne A, Dodd FL, Robertson BC, Forster J, Haskell-Ramsay CF. Multivitamins and minerals modulate whole-body energy metabolism and cerebral blood-flow during cognitive task performance: a double-blind, randomised, placebo-controlled trial. Nutr Metab (Lond). 2016 Feb 11;13:11. doi: 10.1186/s12986-016-0071-4. eCollection 2016. PMID 26870152